CLINICAL TRIAL: NCT03693690
Title: Far Eastern Memorial Hospital
Brief Title: Factors Affecting Therapeutic Efficacy of Vaginal Laser Therapy for Female Stress Urinary Incontinence, and the Effect of Vaginal Laser Therapy on Overactive Bladder Syndrome and Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 107089-F
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Laser Thermotherapy, Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vaginal laser thermotherapy — Laser thermotherapy can increase the stiffness of vaginal wall. It has been reported that vaginal laser therapy can be used to treat stress urinary incontinence.

SUMMARY:
The main aim of this study is to elucidate factors affecting treatment efficacy of vaginal laser therapy.

DETAILED DESCRIPTION:
Laser thermotherapy can increase the stiffness of vaginal wall. It has been reported that vaginal laser therapy can be used to treat stress urinary incontinence. However, factor affecting treatment efficacy of vaginal laser therapy remains unknown. Thus the main aim of this study is to elucidate factors affecting treatment efficacy of vaginal laser therapy. Besides, the durability of vaginal laser therapy will be assessed. The above knowledge should be helpful for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old female
* had stress urinary incontinence symptoms
* Sexual behavior
* No urinary tract infection
* At their own expense for vaginal laser therapy

Exclusion Criteria:

* Abnormal vaginal bleeding
* Vaginal fistula

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Global response assessment | 2 years

SECONDARY OUTCOMES:
Duration of sustained efficacy | 2 years
  Duration of global response assessment ≥ 2 at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, New Taipei City, Banqiao, Taiwan

REFERENCES:
- [Derived] Hsiao SM, Wu WY, Lin HH. Predictors of the efficacy of CO 2 laser therapy for female stress urinary incontinence. J Chin Med Assoc. 2025 Feb 1;88(2):145-150. doi: 10.1097/JCMA.0000000000001193. Epub 2024 Nov 18. PMID 39792642